CLINICAL TRIAL: NCT04419454
Title: Retrospective Evaluation of Cellulite of Laxity Treatment Using Body Tite
Status: Completed | Type: Observational
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DO609568A
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-05

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: BodyTite — retrospectively evaluate this novel treatment approach to improve the appearance of cellulite on the thighs and buttocks by tightening the SFS using RFAL.

SUMMARY:
Retrospective Evaluation of Cellulite of Laxity Treatment Using Body Tite

DETAILED DESCRIPTION:
The purpose of this preliminary report is to retrospectively evaluate this novel treatment approach to improve the appearance of cellulite on the thighs and buttocks by tightening the SFS using RFAL.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18years of age at the time of procedure

  * patients with localized lipodystrophy in the medial or lateral thigh, and visible cellulite of laxity in the lower extremity or buttocks
  * BodyTite treatments performed from January 2018 - May 2019 for Cellulite indication

Exclusion Criteria:

* active infection, collagen disorders, immunocompromised state, medications that mitigate inflammatory response, and propensity for keloid/hypertrophic scaring. o BodyTite treatments performed from March 2018 - May 2019 for lipodystrophy and cellulite of laxity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Sample size will be a result of available charts from a 16-month retrospective review January 2018 - May 2019. The sample will not include any vulnerable populations (pregnant women, minors, or prisoners)
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Photonumeric Cellulite Severity Score | [ Time Frame: Baseline to 6 months posttreatment]
  Change in Photonumeric Cellulite Severity Score 3. Investigator assessment of the cellulite improvement comparing pre and post treatment using Global aesthetic improvement 5-point grading scale (0=No change, 1=1%-24%%, 2=25%-49%, 3=50%-74% improvement, and 4=75%-100%) at all follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Petrs, MD, Principal Investigator
Locations (1):
- Dr. Mark Peters, Germantown, Tennessee, United States